CLINICAL TRIAL: NCT07326436
Title: Comparison of Sympathetic Block Duration and Rebound Sympathetic Activity Rate in Infraclavicular and Supraclavicular Brachial Plexus Blocks Using Perfusion Index and Skin Temperature
Brief Title: Comparison of Sympathetic Blockade Duration in Brachial Plexus Blocks Performed by Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pelin Doğan Uzun, Doctor of medicine, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Brachial Plexus Block
Record Dates: First submitted 2023-04-10; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia, Conduction; Brachial Plexus Blockade; Sympathetic Blockade
Keywords: supraclavicular brachial plexus block; perfusion index; skin temperature; infraclavicular brachial plexus block; sympathetic blockade

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular brachial plexus block (Active Comparator)
  Interventions: Procedure: Supraclavicular brachial plexus block
- Infraclavicular brachial plexus block (Active Comparator)
  Interventions: Procedure: Infraclavicular brachial plexus block

INTERVENTIONS:
Procedure: Supraclavicular brachial plexus block — A linear US probe (7-13 MHz) will be placed in the supraclavicular area in the coronal oblique plane, in-plane technique will be used, and after antisepsis of the area to be blocked, injection will be performed from lateral to medial direction using a 22G 50 mm stimulator needle (Stimuplex A®: B. Braun Melsungen AG, Japan). Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture. A total of 30 mL of 2% prilocaine containing 0.5% bupivacaine and 5 mcg/mL adrenaline in a 1:1 ratio will be used as local anesthetic.
  Arms: Supraclavicular brachial plexus block
Procedure: Infraclavicular brachial plexus block — A linear US probe (7-13 MHz) will be placed in the infraclavicular area through a lateral sagittal approach, in plane technique will be used and injection will be performed using a 22G 100 mm stimulator needle (Stimuplex A®: B. Braun Melsungen AG, Japan) after antisepsis of the area to be blocked. Intermittent negative aspiration will be performed during all procedures to detect possible vascular puncture. A total of 30 mL of 2% prilocaine containing 0.5% bupivacaine and 5 mcg/mL adrenaline in a 1:1 ratio will be used as local anesthetic.
  Arms: Infraclavicular brachial plexus block

SUMMARY:
This prospective comparative study will evaluate the sympathetic effects of ultrasound-guided infraclavicular versus supraclavicular brachial plexus blocks in adults undergoing upper-extremity surgery. Sympathetic tone will be monitored noninvasively with simultaneous bilateral measurements of perfusion index (pulse-oximetry-derived) and skin temperature obtained at baseline and at predefined post-block intervals until return to baseline. The primary outcome is the duration of sympathetic block. Secondary outcomes are between-approach differences in the time course of perfusion index and skin temperature, and the incidence and magnitude of rebound sympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 year old
* ASA I-II
* Patients scheduled for upper extremity surgery
* Fully oriented and able to cooperate
* Patients who signed the informed consent form and gave consent to participate in the study

Exclusion Criteria:

* ASA III-IV-V
* Non-cooperation
* Disease that interferes with sensory block assessment
* Known allergy to the medicines to be used
* Pregnant patients
* Coagulopathy or thrombocytopenia
* Patients with anatomical abnormalities or active infection at the points of application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
Difference in duration of sympathetic blockade after different US-guided brachial plexus blocks | Twenty-four hours after nerve blockage

SECONDARY OUTCOMES:
Change in perfusion index between infraclavicular and supraclavicular approaches | Twenty-four hours after nerve blockage
  The perfusion index measured by pulse oximetry will be recorded at baseline and twenty-four hours after brachial plexus block. The outcome measure is defined as the change in perfusion index value between the two time points and compared between block approaches.

CONTACTS AND LOCATIONS:
Locations (1):
- Bozyaka Training and Research Hospital, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided